CLINICAL TRIAL: NCT06055907
Title: Anti-Xa Activity in Patients Receiving Different Vasopressors.
Brief Title: Influence of Vasopressors on Anti-Xa Activity in Critically Ill Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Sponsor
Other Study IDs: SKN+JS
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Critical Illness; Thrombosis
MeSH Terms: conditions — Critical Illness; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NOR+ARG: Critically ill patients receiving norepinephrine and argipressin, with antithrombotic prophylaxis with 5000 IU of dalteparin.
  Interventions: Diagnostic Test: Serum anti-Xa activity
- NOR: Critically ill patients receiving norepinephrine alone, with antithrombotic prophylaxis with 5000 IU of dalteparin.
  Interventions: Diagnostic Test: Serum anti-Xa activity

INTERVENTIONS:
Diagnostic Test: Serum anti-Xa activity — 4 hours after third dose of dalteparin, serum anti-Xa activity is measured

SUMMARY:
Critically ill patients require antithrombotic prophylaxis. At the same time, majority of them is receiving various vasopressors. The aim of the study is to determine whether there is a difference in anti-Xa activity, which is a marker of anti thrombotic activity of low molecular weight heparins, between the patients receiving norepinephrine with argipressin, compared to those receiving norepinephrine alone.

ELIGIBILITY:
Inclusion Criteria:

* Circulatory failure
* Supported by continuous infusion of noradrenaline or noradrenaline and argipressin
* Receiving subcutaneous dalteparin for the prevention of venous thromboembolism.

Exclusion Criteria:

* Contraindications for dalteparin
* Severe coagulopathy
* Acute or subacute bacterial endocarditis
* Pregnant women
* BMI (body mass index) > 30kg/m2
* Chronic kidney disease with eGFR (estimated glomerular filtration rate) < 30 ml/min/1.73 m2
* Renal replacement therapy
* The patient died within 52 hours of starting VTE (venous thromboembolism) prophylaxis with dalteparin

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohort study will be conducted on a population of 50 adult patients of both sexes treated in the Intensive Care Unit at the University Clinical Center in Gdansk, Poland.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Anti-Xa activity | 4 hours after third dose
  IU anty-Xa/ml

CONTACTS AND LOCATIONS:
Overall Officials: Radosław Owczuk, MD., PhD., Prof., Study Director — Medical University of Gdansk
Locations (1):
- Medical University of Gdańsk - Departament of Anesthesiology and Intensive Care, Gdansk, Poland